CLINICAL TRIAL: NCT00885924
Title: Desmopressin as Treatment for Postoperative Bleeding After Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: to include required number of patients took too much time
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4.2008.947
Record Dates: First submitted 2009-04-02; First posted 2009-04-22 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Hemorrhage; Postoperative Blood Loss
Keywords: postoperative Hemorrhage; Hemorrhage; Vasopressin; Blood Loss, Surgical
MeSH Terms: conditions — Hemorrhage; Postoperative Hemorrhage; Diabetes Insipidus; Blood Loss, Surgical | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Active Comparator): Desmopressin 0.3 microgram/kg
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): NaCl 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — Desmopressin 0.3 microgram/kg as an intravenous infusion given during 20 min.
  Other Names: Octostim, Ferring ATC-nr.:H01B A02
  Arms: Active treatment
Drug: Placebo — NaCl 0.9%
  Arms: Placebo

SUMMARY:
Some patients undergoing cardiac surgery develop excessive postoperative bleeding. Cardiopulmonary bypass causes platelet dysfunction. Several studies have documented the ability of desmopressin to reduce hemorrhage in a variety of congenital and acquired platelet disorders. In this study the investigators will investigate wether desmopressin reduces postoperative microvascular bleeding. The investigators will investigate wether desmopressin reduces platelet activation as measured by plasma concentration of neutrophil activating peptid 2 and by flow cytometry. The primary endpoint of the study will, however, be total postoperative bleeding and need for transfusions of blood components after surgery. The need for transfusions will be registered during the whole hospital stay. Patient with excessive postoperative bleeding (more than 250 ml for one hour, or more than 150ml for two hours during the first four hours) will be randomized into two groups and given either desmopressin or placebo (0,9% sodium chloride) as an intravenous infusion. Blood samples for plasma concentration measurements will be drawn before infusion of desmopressin/placebo, immediately after the infusion and 20 hours postoperatively. Postoperative bleeding will be registered for 16 hours. The need for any transfusions of blood products will be registered for the whole hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age scheduled for cardiac surgery
* Excessive postoperative bleeding, more than 250 ml for one hour, or more than 150ml for two hours during the first four hours

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with a medical condition known to influence the hemostatic system
* Patients treated with clopidogrel or systemic steroids during the last week before surgery
* Patients with INR above 1.5
* Patients who are not able to give written informed concent
* Unstable patients who need other transfusion limits than in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Transfusion of blood components | During postoperative stay

SECONDARY OUTCOMES:
Postoperative hemorrhage | First 16 hours postoperatively
Platelet activation | 20 hours postoperatively
Activation of coagulation | 20 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Guri Greiff, MD, Principal Investigator — StOalvs Hospital
Locations (1):
- StOlavs Hopital, Trondheim, Trondheim, Norway